CLINICAL TRIAL: NCT00234585
Title: A Prospective Randomized Multicenter Study Comparing the Safety and Efficacy of Renal Artery Stenting With/Without Distal Protection Device (AngioGuard) and With/Without the Use of a Platelet Aggregator Inhibitor (Abciximab-Reopro) (RESIST)
Brief Title: Prospective Randomized Study Comparing Renal Artery Stenting (RESIST)With/Without Distal Protection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toledo Health Science Campus (Other)
Collaborators: Centocor, Inc. (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xMUO-01
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Renal Artery Stenosis
MeSH Terms: conditions — Renal Artery Obstruction

INTERVENTIONS:
Device: Renal Artery Stent with Protective Device/Drug

SUMMARY:
This study is designed to demonstrate the safety and efficacy of using a protective device/drug to prevent renal injury during renal artery stenting and to assess whether the preventative effects are measurable and if there is a differential treatment effect for either device alone or in combination.

DETAILED DESCRIPTION:
This study is designed to demonstrate the safety and efficacy of using protective device/drug to prevent renal injury during renal artery stenting (RAS) and to assess whether the preventative effects are measurable, and if there is a differential treatment effect for either device alone or in combination.

Specific goals of the study include:

* To establish device and drug safety
* To identify appropriate markers for renal injury
* To measure effectiveness of drug and device
* To enable the design of FDA efficacy trials for renal artery stenting inclusive of device and or drug

The study will address the four following hypotheses:

* AngioGuard™ distal protection device provides significant protection from atheroembolization during RAS procedures as measured by affected kidney GFR at 1 month after the procedure.
* Abciximab (ReoPro) offers protection against platelet aggregation and embolization as measured by affected kidney GFR at 1 month after the procedure.
* AngioGuard™ and Abciximab are safe, alone and in combination.
* Is there an interaction effect between AngioGuard™ and ReoPro for efficacy and safety?

ELIGIBILITY:
Inclusion Criteria:

Any one or more of the following:

Meet Angiographic criteria plus

* Systemic hypertension at baseline, or a history of hypertension
* Congestive heart failure at baseline, or a history of CHF
* Renal insufficiency at baseline, or a history of renal insufficiency
* Angina, or a history of angina

Exclusion Criteria:

* Less than 18 years old
* Contraindications to device/drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-08; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Glomerular Filtration Rate
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cooper, M.D., Principal Investigator — Medical University of Ohio
Locations (1):
- Medical University of Ohio, Toledo, Ohio, United States

REFERENCES:
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730
- [Derived] Yu H, Zhang D, Haller S, Kanjwal K, Colyer W, Brewster P, Steffes M, Shapiro JI, Cooper CJ. Determinants of renal function in patients with renal artery stenosis. Vasc Med. 2011 Oct;16(5):331-8. doi: 10.1177/1358863X11419998. Epub 2011 Sep 9. PMID 21908683
- [Derived] Tian J, Haller S, Periyasamy S, Brewster P, Zhang H, Adlakha S, Fedorova OV, Xie ZJ, Bagrov AY, Shapiro JI, Cooper CJ. Renal ischemia regulates marinobufagenin release in humans. Hypertension. 2010 Nov;56(5):914-9. doi: 10.1161/HYPERTENSIONAHA.110.155564. Epub 2010 Sep 7. PMID 20823380
- [Derived] Kanjwal K, Cooper CJ, Virmani R, Haller S, Shapiro JI, Burket MW, Steffes M, Brewster P, Zhang H, Colyer WR Jr. Predictors of embolization during protected renal artery angioplasty and stenting: Role of antiplatelet therapy. Catheter Cardiovasc Interv. 2010 Jul 1;76(1):16-23. doi: 10.1002/ccd.22469. PMID 20209644
- [Derived] Kanjwal K, Haller S, Steffes M, Virmani R, Shapiro JI, Burket MW, Cooper CJ, Colyer WR Jr. Complete versus partial distal embolic protection during renal artery stenting. Catheter Cardiovasc Interv. 2009 May 1;73(6):725-30. doi: 10.1002/ccd.21932. PMID 19198007
- [Derived] Cooper CJ, Haller ST, Colyer W, Steffes M, Burket MW, Thomas WJ, Safian R, Reddy B, Brewster P, Ankenbrandt MA, Virmani R, Dippel E, Rocha-Singh K, Murphy TP, Kennedy DJ, Shapiro JI, D'Agostino RD, Pencina MJ, Khuder S. Embolic protection and platelet inhibition during renal artery stenting. Circulation. 2008 May 27;117(21):2752-60. doi: 10.1161/CIRCULATIONAHA.107.730259. Epub 2008 May 19. PMID 18490527